CLINICAL TRIAL: NCT02149355
Title: Teeth and Jaw Misalignment in Patients Suffering From Congenital Fourth Cranial Nerve Palsy
Acronym: IVPareseZahn
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH 2013-0342; KEK-ZH 2013-0342 (Other: cantonal ethical committee Zurich)
Record Dates: First submitted 2014-04-07; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Fourth Cranial Nerve Palsy
Keywords: teeth position; jaw alignment
MeSH Terms: conditions — Trochlear Nerve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- controls: teeth molding in subjects without congenital fourth nerve palsy
  Interventions: Other: teeth molding
- congenital fourth nerve palsy: teeth molding in patients suffering from congenital fourth nerve palsy
  Interventions: Other: teeth molding

INTERVENTIONS:
Other: teeth molding — teeth molding in patients suffering from congenital fourth nerve palsy

SUMMARY:
Patients suffering from congenital fourth cranial nerve palsy may have misalignment of jaws as well as teeth due to head tilt in childhood.

DETAILED DESCRIPTION:
Measurement of teeth and jaw parameters in patients suffering from congenital fourth cranial nerve palsy compared to patients without fourth cranial nerve palsy.

ELIGIBILITY:
Inclusion Criteria:

* unilateral congenital fourth nerve palsy
* natural teeth occlusion
* age > 18 years

Exclusion Criteria:

* bilateral fourth nerve palsy
* no natural teeth occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients suffering from congenital fourth nerve palsy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
angle between teeth positions from upper and lower jaw | 3 to 6 months after recruitment
  The angle between teeth positions from upper and lower jaw will be measured using teeth molding.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Landau, Prof MD, Study Chair — University Hospital Zurich, ophthalmology department
Locations (1):
- UniversityHospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- See also: official homepage of swiss federal government — http://www.kofam.ch